CLINICAL TRIAL: NCT04849078
Title: Translation of Dizziness Handicap Inventory Scale Into Local Languages of Pakistan
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00958 Sidra Ali Naqvi
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Vertigo; Dizziness
Keywords: vertigo; dizziness; dizziness handicap inventory
MeSH Terms: conditions — Vertigo; Dizziness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the present study is to translate the Dizziness Handicap Inventory Scale into Urdu, Pashto, Punjabi, Sindhi and Balochi languages. Along with validation of the translated versions by evaluating their validity and reliability in the people of Pakistan, speaking respective languages and suffering from vertigo and dizziness. No such study has been previously conducted in the Pakistan region which translates the scale and follows the proper cross-culture adaptation.

DETAILED DESCRIPTION:
Dizziness is one of the most common symptoms of many diseases that not only affects the daily activities of the patient but also negatively alters their jobs and functions. Moreover, mostly the patients having dizziness due to vestibular causes are known to face more problems as compared to the others. A precisely valid and reliable tool has been already designed for the measurement of dizziness while keeping the common complaints of patients in mind. The dizziness handicap inventory (DHI) was introduced in 1990 by Jacobson and Newman. The mentioned questionnaire comprises 25 questions that categorize the dizziness effects in three main areas namely; functional (9 questions, 36 points), emotional (9 questions, 36 points) and physical (7 questions, 28 points). The maximum score is 100 and the minimum is 0. The higher the score, the greater handicap is considered. It has high internal consistency. This tool is widely used in clinical setups to evaluate the condition of the patients and determine the levels to which their quality of life has been affected by dizziness. Additionally, it is very easy to be filled and hardly takes 10 minutes at maximum. The DHI is highly compatible with the international classification of functioning, disability and health tool, which was standardized by WHO in 2001 for measuring the effects of various diseases. The aim of DHI is to evaluate the self-perceived handicap effects of dizziness. The target population are the patients suffering from dizziness due to brain injuries, multiple sclerosis and vestibular disorders.

Since 1990, the DHI has been translated into various languages in order to make its application better. Some examples of the translated languages include Arabic, Brazilian, Spanish, Chinese, Italian, Dutch, French, Norwegian, and German. All of these translated versions have been proved to be very useful, with high validity, reliability and internal consistency.

Thus, The DHI is considered the most beneficial questionnaire for the evaluation of dizziness and unsteadiness, especially related to vestibular rehabilitation. However, this questionnaire does not have any versions that can be utilized in Pakistan such as Urdu, Pushto, Punjabi, Sindhi and Balochi. The purpose of this study is to translate the DHI into Urdu, Pushto, Punjabi, Sindhi and Balochi languages and then evaluating the validity and reliability of these versions in order to make this questionnaire available for research and clinics for the population of Pakistan.

ELIGIBILITY:
Inclusion Criteria:

* The patient suffering from vertigo and dizziness for at least 1 month and
* The ability to walk independently or do their routine tasks will be included in the study.
* Patients should be capable to complete the questionnaire without any help.

Exclusion Criteria:

* Patients suffering from blindness,
* musculoskeletal abnormalities,
* neurologic disorder, or paralysis in ENT or neurologic evaluation by ENT and
* neurologist will be excluded from the study.
* Also, if the patients are unable to cooperate then, they will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To meet inclusion criteria participants diagnosed with dizziness and vertigo, clinically stable, and able to read the local language version of the Dizziness Handicap Inventory. Then patient response will be checked on the translated versions
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cross-Cultural Translation of Dizziness Handicap Inventory Scale into the local languages (Punjabi, Pashto, Sindhi, Balochi and Urdu) | 6 months
  The Dizziness Handicap Inventory Scale is a first-hand measure of disability for patients with vertigo and dizziness. The mentioned questionnaire comprises 25 questions that categorize the dizziness effects in three main areas namely; functional (9 questions, 36 points), emotional (9 questions, 36 points) and physical (7 questions, 28 points). The maximum score is 100 and the minimum is 0. The higher the score, the greater handicap is considered. It distinguishes itself from other published scales as it has an approach that deals with the concepts of disability and its assessment. Its translation is to be done in the local languages of Pakistan through a rigorous and approved process.

SECONDARY OUTCOMES:
Reliability of translated versions | 6 months
  To determine the reliability of cross-culturally adapted and the translated Dizziness Handicap Inventory versions in patients with vertigo and dizziness of respective languages۔ Reliability or reproducibility refers to the ability of a measure to produce the same results when administered at two or more interval between different visits of the patient. Thus this will be measured through test re-test reliability.
Validity of translated versions | 6 months
  To determine the validity of cross-culturally adapted and the translated Dizziness Handicap Inventory versions in patients with vertigo and dizziness of respective languages۔ Validity is how accurate the results are. Thus this will be measured through various parameters to validate the translated versions as appropriate and applicable.

CONTACTS AND LOCATIONS:
Overall Officials: Imran Amjad, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Fedral, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Poon DM, Chow LC, Au DK, Hui Y, Leung MC. Translation of the dizziness handicap inventory into Chinese, validation of it, and evaluation of the quality of life of patients with chronic dizziness. Ann Otol Rhinol Laryngol. 2004 Dec;113(12):1006-11. doi: 10.1177/000348940411301212. PMID 15633905
- [Background] Nola G, Mostardini C, Salvi C, Ercolani AP, Ralli G. Validity of Italian adaptation of the Dizziness Handicap Inventory (DHI) and evaluation of the quality of life in patients with acute dizziness. Acta Otorhinolaryngol Ital. 2010 Aug;30(4):190. PMID 21253284
- [Background] Kurre A, Bastiaenen CH, van Gool CJ, Gloor-Juzi T, de Bruin ED, Straumann D. Exploratory factor analysis of the Dizziness Handicap Inventory (German version). BMC Ear Nose Throat Disord. 2010 Mar 15;10:3. doi: 10.1186/1472-6815-10-3. PMID 20230621
- [Background] Alsanosi AA. Adaptation of the dizziness handicap inventory for use in the Arab population. Neurosciences (Riyadh). 2012 Apr;17(2):139-44. PMID 22465888
- [Background] Castro AS, Gazzola JM, Natour J, Gananca FF. [Brazilian version of the dizziness handicap inventory]. Pro Fono. 2007 Jan-Apr;19(1):97-104. doi: 10.1590/s0104-56872007000100011. Portuguese. PMID 17461352
- [Background] Perez N, Garmendia I, Martin E, Garcia-Tapia R. [Cultural adaptation of 2 questionnaires for health measurement in patients with vertigo]. Acta Otorrinolaringol Esp. 2000 Oct;51(7):572-80. Spanish. PMID 11270034
- [Background] Vereeck L, Truijen S, Wuyts F, Van de Heyning PH. Test-retest reliability of the Dutch version of the Dizziness Handicap Inventory. B-ENT. 2006;2(2):75-80. PMID 16910291
- [Background] Nyabenda A, Briart C, Deggouj N, Gersdorff M. [Normative study and reliability of French version of the dizziness handicap inventory]. Ann Readapt Med Phys. 2004 Apr;47(3):105-13. doi: 10.1016/j.annrmp.2003.11.002. French. PMID 15059673
- [Background] Tamber AL, Wilhelmsen KT, Strand LI. Measurement properties of the Dizziness Handicap Inventory by cross-sectional and longitudinal designs. Health Qual Life Outcomes. 2009 Dec 21;7:101. doi: 10.1186/1477-7525-7-101. PMID 20025754
- [Background] Kurre A, van Gool CJ, Bastiaenen CH, Gloor-Juzi T, Straumann D, de Bruin ED. Translation, cross-cultural adaptation and reliability of the german version of the dizziness handicap inventory. Otol Neurotol. 2009 Apr;30(3):359-67. doi: 10.1097/MAO.0b013e3181977e09. PMID 19225437